CLINICAL TRIAL: NCT01942824
Title: Adult Influenza Vaccination Text Message Reminders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAK5058_2
Record Dates: First submitted 2013-09-08; First posted 2013-09-16 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Text Message
  Interventions: Behavioral: Text Messages
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Text Messages
  Arms: Intervention

SUMMARY:
Influenza infection leads to on average 24,0000 deaths and 150,000 hospitalizations annually. While vaccination is the cornerstone of preventing influenza infection, vaccination coverage in adults is low with only 35% vaccinated by end of November. Latino adults have the lowest coverage rates. Text message reminders have been used successfully for improving influenza vaccination for children. This study will assess the use of text messaging to improve influenza vaccination coverage rates in a largely minority, publicly insured adult population.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age,
* at least one visit to the AIM clinic during the previous year
* a cell phone number in the registration system
* fluent in English or Spanish. Exclusion criteria

Exclusion Criteria:

- Receipt of influenza vaccination during the 2013-2014 influenza season prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7250 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Timeliness of vaccination | 6 months
  Days from start of intervention to vaccination

SECONDARY OUTCOMES:
Receipt of influenza vaccine dose | 15 weeks
  Proportion of individuals in each group receiving an influenza dose by December 31, 2013
Receipt of Influenza vaccine dose, end of season | 28 weeks
  Proportion of individuals in each group receiving an influenza dose by March 31st, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Steven Shea, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States